CLINICAL TRIAL: NCT01906346
Title: Impact of a Non-Drug Choice on Cocaine Reinforcement
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Joshua A. Lile, Ph.D. (Other)
Responsible Party: Sponsor-Investigator, Joshua A. Lile, Ph.D., Joshua A. Lile, Ph.D., Associate Professor of Behavioral Science, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: R01DA033364-01 (NIH)
Record Dates: First submitted 2013-07-16; First posted 2013-07-24 (Estimated); Results first posted 2019-05-17 (Actual); Last update posted 2019-05-17 (Actual); Status verified 2019-04

CONDITIONS: Cocaine Dependence
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Cocaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Low Value Alternative Reinforcer (Experimental): A low value reinforcer will be made available as an alternative to cocaine and placebo.
  Interventions: Drug: Cocaine; Drug: Placebo
- Medium Value Reinforcer (Experimental): A medium value reinforcer will be made available as an alternative to cocaine and placebo.
  Interventions: Drug: Cocaine; Drug: Placebo
- High Value Reinforcer (Experimental): A high value reinforcer will be made available as an alternative to cocaine and placebo.
  Interventions: Drug: Cocaine; Drug: Placebo

INTERVENTIONS:
Drug: Cocaine — Three active doses of cocaine will be made available for self-administration during experimental sessions.
Drug: Placebo — Placebo cocaine will be made available for self-administration during experimental sessions.

SUMMARY:
Cocaine-use disorders continue to be a significant public health concern, yet no effective medications have been identified. The goal of this study is to establish a research platform for the development of medications for treatment of cocaine abuse and dependence. This study will incorporate self-administration procedures and a non-drug alternative reinforcer, which is hypothesized to reduce the reinforcing effects of cocaine.

ELIGIBILITY:
Inclusion Criteria:

* Cocaine dependence, otherwise healthy

Exclusion Criteria:

* Laboratory results outside of clinically acceptable ranges, history of or current serious physical or psychiatric disease

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2014-01; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joshua A Lile, Ph.D, Principal Investigator — University of Kentucky
Locations (1):
- Laboratory of Human Behavioral Pharmacology, Lexington, Kentucky, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Randomized Combination of One Drug Dose and One Money Value: Low, medium and high value monetary reinforcers are made available as an alternative to cocaine and placebo during experimental sessions.
  Cocaine: Three active doses of cocaine are made available for self-administration during experimental sessions.
  Placebo: Placebo cocaine is made available for self-administration during experimental sessions.
Period: Overall Study
Arm/Group | Randomized Combination of One Drug Dose and One Money Value
Started | 9
Completed | 8
Not Completed | 1
Not completed — AEs | 1

BASELINE CHARACTERISTICS:
Arm/Group | Randomized Combination of One Drug Dose and One Money Value
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: The Number of Times Cocaine Was Selected in the Presence of a Monetary Reward Alternative
Description: The reinforcing effects of cocaine were determined using a modified progressive ratio procedure in which subjects made 9 choices between each available cocaine dose and one of three money alternatives.
Time Frame: 9 choice trials per cocaine dose level with each trial separated by 30 minutes
Measure: Mean (Standard Error); unit: cocaine choices
Groups:
- Low Value Alternative Reinforcer: A low value reinforcer was made available as an alternative to cocaine and placebo.
  Cocaine: Three active doses of cocaine will be made available for self-administration during experimental sessions.
  Placebo: Placebo cocaine will be made available for self-administration during experimental sessions.
- Medium Value Reinforcer: A medium value reinforcer was made available as an alternative to cocaine and placebo.
  Cocaine: Three active doses of cocaine will be made available for self-administration during experimental sessions.
  Placebo: Placebo cocaine will be made available for self-administration during experimental sessions.
- High Value Reinforcer: A high value reinforcer was made available as an alternative to cocaine and placebo.
  Cocaine: Three active doses of cocaine will be made available for self-administration during experimental sessions.
  Placebo: Placebo cocaine will be made available for self-administration during experimental sessions.
Arm/Group | Low Value Alternative Reinforcer | Medium Value Reinforcer | High Value Reinforcer
Number analyzed (Participants) | 8 | 8 | 8
cocaine choices
  Placebo Cocaine | 2.75 (1.39) | 1.38 (0.53) | 1.38 (0.53)
  3 mg/70 kg Cocaine | 4.75 (1.24) | 5.88 (1.17) | 4.00 (1.52)
  10 mg/70 kg Cocaine | 7.38 (1.07) | 6.13 (1.47) | 6.38 (1.41)
  30 mg/70kg Cocaine | 7.63 (1.12) | 7.13 (1.13) | 6.38 (1.22)

ADVERSE EVENTS:
Time Frame: 15 days per subject.
Description: Adverse event reporting consists of each experimental session in which a single cocaine dose and monetary reinforcer were available as choice alternatives, as well as during the conduct of a medical safety session in which cocaine doses are administered prior to choice sessions.
Arm/Group | Randomized Combination of One Drug Dose and One Money Value
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 1/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Randomized Combination of One Drug Dose and One Money Value (N=9)
Nausea and vomiting (Gastrointestinal disorders) | 1 (3) — Three incidents of nausea and vomiting that did not coincide with drug administration.
Difficulty obtaining IV line (Investigations) | 1 — Multiple sticks required to place IV catheter

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No